CLINICAL TRIAL: NCT05583812
Title: A Double-Blinded, Randomized, and Placebo-Controlled Phase 1 Study to Assess the Safety, Tolerability and Pharmacokinetics Profile of Single and Multiple Ascending Doses of FB2001 for Inhalation in Healthy Chinese Adults
Brief Title: A Study of FB2001 for Inhalation in Healthy Chinese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Frontier Biotechnologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FB2001-103
Record Dates: First submitted 2022-10-08; First posted 2022-10-18 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-09

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — FB2001; Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SAD Dose 1 (Experimental): Subjects will receive FB2001 or placebo for inhalation once on DAY 1
  Interventions: Drug: FB2001 for inhalation; Drug: FB2001 for inhalation placebo
- SAD Dose 2 (Experimental): Subjects will receive FB2001 or placebo for inhalation once on DAY 1
  Interventions: Drug: FB2001 for inhalation; Drug: FB2001 for inhalation placebo
- MAD Dose 1 (Experimental): Subjects will receive FB2001 or placebo for inhalation twice daily during the dosing period
  Interventions: Drug: FB2001 for inhalation; Drug: FB2001 for inhalation placebo
- MAD Dose 2 (Experimental): Subjects will receive FB2001 or placebo for inhalation twice daily during the dosing period
  Interventions: Drug: FB2001 for inhalation; Drug: FB2001 for inhalation placebo

INTERVENTIONS:
Drug: FB2001 for inhalation — FB2001 once or twice daily inhalation
  Other Names: DC402234
Drug: FB2001 for inhalation placebo — FB2001 placebo once or twice daily inhalation

SUMMARY:
FB2001 is a novel inhalable preparation being developed for COVID-19 treatment. A Double-Blinded, Randomized, and Placebo-Controlled Phase 1 Study to Assess the Safety, Tolerability and Pharmacokinetics Profile of Single and Multiple Ascending Doses of FB2001 in Healthy Chinese Adults

DETAILED DESCRIPTION:
Coronaviruses belong to the genus of coronavirus of the family coronaviruses. The viruses of the coronavirus genus are positive-sense single-stranded RNA viruses with envelopes, which are approximately 80-160 nm in diameter. Their genetic material is the largest among all RNA viruses and can infect both humans and animals. Coronaviruses can cause respiratory, intestinal, hepatic, and nervous system diseases of different severities. A total of 7 coronaviruses have been found, in which HCoV-229E, HCoV-OC43, HCoV-NL63 and HCoV-HKU1 mainly lead to mild and self-limiting upper respiratory tract infections in infected humans, such as common cold; two new types of β-coronaviruses have emerged in the past 12 years, namely severe acute respiratory syndrome (SARS-CoV) and Middle East respiratory syndrome (MERS-CoV), and these two viruses can cause severe human diseases.

This is a Phase 1, randomized, double-blinded, placebo controlled, dose escalation study of FB2001 in healthy adult volunteers.The study aims to evaluate the safety, tolerability and pharmacokinetic profile of FB2001 administered by aerosol inhalation after single and multiple ascending doses.Approximately 32 participants will be sequentially enrolled into either 1 of 2 SAD cohorts (n=8 per cohort), or 1 of 2 MAD cohorts (n= 8 per cohort). An adaptive dose escalation schedule will be employed for both SAD and MAD parts of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese male and female volunteers aged 18 to 60 years (including the threshold);
2. Male weight ≥ 50 kg and female weight ≥ 45 kg with body mass index (BMI) = weight (kg)/height2 (m2) BMI within the range of 19 to 26 kg/m2 (including the threshold);
3. Voluntary participation in the trial and full understanding of the trial content, process and possible adverse effects;
4. Willing to cooperate and be able to participate in the study, comply with all requirements of the program, and sign informed consent.

Exclusion Criteria:

1. Participation in any clinical trial within 3 months prior to the administration of the drug;
2. Previous history of respiratory disease such as acute exacerbation of chronic obstructive pulmonary disease, pulmonary fibrosis, pulmonary hypertension, pulmonary oedema, interstitial lung lesions, bronchial asthma, paradoxical bronchospasm, or pharyngeal ulceration, oedema, or previous pharyngeal, tracheal/bronchial and pulmonary surgery which the investigator considers to be clinically significant;
3. A history of cardiovascular, endocrine, neurological, digestive, genitourinary, haematological, immunological (including personal or family history of hereditary immunodeficiency), or metabolic abnormalities which the investigator considers to be clinically significant;
4. Volunteers with a history of allergy to the product and excipients, or a history of hypersensitivity to drugs, foods or other substances;
5. Volunteers with a history of intolerance to venipuncture or needle phobia and bloodsickness；
6. Volunteers who have undergone surgery within 6 months prior to dosing which in the judgment of the investigator would interfere with the absorption, distribution, metabolism, or excretion, or who have undergone or are scheduled to undergo surgery during the study period within 4 weeks prior to dosing；
7. Volunteers having used any medication (including prescription, over-the-counter, herbal, nutraceuticals, etc.) within 14 days prior to administration of the experimental drug；
8. volunteers having used any drug metabolism inhibitors or inducers within 30 days prior to the administration of the drug；
9. Volunteers receiving a vaccine or attenuated vaccine within 14 days prior to dosing, or planning to have a vaccine administered during the trial；
10. Volunteers having donated or lost blood (>400 mL) within 3 months prior to drug administration or intending to donate blood or blood components during or up to 3 months after the end of the trial；
11. substance abusers or having used drugs within 1 year prior to dosing；
12. smokers, or unable to stop using any tobacco-based products during the trial；
13. alcoholics or regular drinkers of alcohol within 6 months prior to the administration；
14. Volunteers consuming excessive amounts of tea, coffee and/or caffeinated beverages on a daily basis or requiring continued drinking during the trial；
15. volunteers having ingested food within 7 days prior to administration that may interfere with the metabolism of the drug in vivo or will be unwilling to stop consuming these foods during the trial.
16. Volunteers with special dietary requirements unable to comply with a uniform diet.
17. volunteers (or their partners) planning to pregnant，donating sperm and oocytes or unwilling to use one or more non-pharmaceutical contraceptive measures within the period of the trial and up to 3 months after the trial ；
18. Female volunteers are pregnant or lactating; or are having unprotected sex within 2 weeks prior to administration; or are using oral contraceptives within 30 days prior to the administration or using long-acting estrogen or progestin injections or implant tablets within 6 months prior to administration；
19. volunteers with clinically significant abnormalities in physical examination, 12-lead ECG, vital signs (blood pressure, pulse, temperature, SpO2), chest X-ray, pregnancy tests, laboratory tests, pulmonary function tests；
20. Pulmonary function tests: those with FEV1 measured/FEV1 expected ≤ 80% or FVC ≤ 80% of the expected value；
21. Positive Niacin test result.
22. Positive drug test result.
23. positive alcohol breath test.
24. inability to use the nebulizer device correctly or failure of training in inhalant administration.
25. The volunteer may be unable to complete the study for other reasons or has other reasons judged by the investigator as inappropriate for participation in the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability after single and multiple doses of FB2001 in healthy subjects | Day 7 or Day 14
  Assessment of safety by monitoring the incidence of AE after drug administration
Pharmacokinetic parameter (AUC0-t) | Day 7 or Day 14
  Pharmacokinetic outcome measures: Estimate of steady state AUC0-t for single and multiple dose administration of FB2001 for Inhalation
Pharmacokinetic parameter (Cmax) | Day 7 or Day 14
  Pharmacokinetic outcome measures: Estimate of steady state Cmax for single and multiple dose administration of FB2001 for Inhalation

CONTACTS AND LOCATIONS:
Overall Officials: Xin Li, PhD, Principal Investigator — The Third Hospital of Changsha
Locations (1):
- The Third Hospital of Changsha, Changsha, China